CLINICAL TRIAL: NCT02374073
Title: Effectiveness of Functional Massage of the Teres Major Muscle in Patients With Subacromial Impingement Syndrome. A Randomized Controlled Pilot Study
Brief Title: Functional Massage of Teres Major Muscle
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P13/082
Record Dates: First submitted 2015-02-12; First posted 2015-02-27 (Estimated); Last update posted 2015-02-27 (Estimated); Status verified 2015-02

CONDITIONS: Subacromial Impingement Syndrome; Trigger Points
MeSH Terms: conditions — Shoulder Impingement Syndrome

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group (Experimental): Treated with protocolized physiotherapy and functional massage
  Interventions: Other: Functional Massage; Other: Protocolized physiotherapy
- Control group (Experimental): Treated with protocolized physiotherapy
  Interventions: Other: Protocolized physiotherapy

INTERVENTIONS:
Other: Functional Massage — The functional massage is a manual therapy technique, indicated in cases of painful muscle tightness that combines a rhythmical and non painful passive joint mobilization in the direction of muscle stretching together with compression/decompression of the muscle to be treated.
  Arms: Intervention group
Other: Protocolized physiotherapy — therapeutic exercises, analgesic electrotherapy and cryotherapy

SUMMARY:
Purpose: Subacromial impingement syndrome is the most common shoulder condition. Myofascial trigger points in teres major muscle can be associated with this syndrome. The investigators objective is to find out if adding manual therapy specifically for teres major trigger points can produce better results in these patients.

Method: A randomized controlled pilot study was carried out. Fifty people were randomly assigned to one of two groups: intervention group or control group. Both groups received a protocolized physical therapy treatment while the intervention group additionally received manual therapy for teres major trigger points.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and over
* Clinical diagnosis of Subacromial Impingement Syndrome.
* Detectable trigger points in teres major muscle.
* Sign informed consent form.

Exclusion Criteria:

* Presence of wounds or cutaneous alterations in the shoulder region
* Previous surgery in the shoulder
* Presence of acute inflammatory process in the shoulder (< 7 days),
* Being involved in litigation or compensation processes
* Not having a domain of the language that could make the informed consent not understandable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2014-01; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Change in Pain Intensity (visual analogue scale) | Change from baseline to 3 weeks
  Using a Visual analogue scale

SECONDARY OUTCOMES:
Change in Function (Abbreviated Constant-Murley score) | Change from baseline to 3 weeks
  Using the Abbreviated Constant-Murley score
Change in Active Range of Motion | Change from baseline to 3 weeks
  Flexion, extension, abduction, external rotation and internal rotation